CLINICAL TRIAL: NCT06495190
Title: Age-related Cognitive Changes: Effects of Combined Flavonoid Intake and Physical Exertion Mediated by the Gut Microbiome
Brief Title: Cognition, Flavonoids, Exercise, Gut Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HS-24-27
Record Dates: First submitted 2024-07-03; First posted 2024-07-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Cognitive Decline, Mild
Keywords: aging; flavonoids; exercise; gut microbiome
MeSH Terms: conditions — Cognitive Dysfunction; Lymphoma, Follicular; Motor Activity | interventions — blueberry extract; Walking

STUDY DESIGN:
Intervention Model Description: This study will employ a randomized, double-blind, placebo controlled, parallel research design, with participants assigned to one of 4 arms for the 12-week trial period: 1) blueberry + walking; blueberry + stretching; placebo + walking; placebo + stretching.
Who Masked: Participant, Investigator
Masking Description: Investigators and study participants will be blind to treatment allocation, with the blueberry and placebo supplements administered in identical packets.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Blueberry + walking (Experimental): Blueberry intake combined with walking exercise.
  Interventions: Dietary Supplement: Blueberry; Behavioral: Walking
- Blueberry + stretching (Experimental): Blueberry intake combined with stretching exercise.
  Interventions: Dietary Supplement: Blueberry; Behavioral: Stretching
- Placebo + walking (Active Comparator): Placebo intake combined with walking exercise.
  Interventions: Behavioral: Walking; Dietary Supplement: Placebo
- Placebo + stretching (Active Comparator): Placebo intake combined with stretching exercise.
  Interventions: Dietary Supplement: Placebo; Behavioral: Stretching

INTERVENTIONS:
Dietary Supplement: Blueberry — 50 g/d blueberry powder supplement
  Arms: Blueberry + stretching; Blueberry + walking
Behavioral: Walking — Five 45-min walking sessions per week
  Other Names: Stretching
  Arms: Blueberry + walking; Placebo + walking
Dietary Supplement: Placebo — 50 g/d placebo powder supplement
  Arms: Placebo + stretching; Placebo + walking
Behavioral: Stretching — Five 45-min stretching sessions per week
  Arms: Blueberry + stretching; Placebo + stretching

SUMMARY:
This NIH project will examine the effects of routine flavonoid-rich blueberry intake (12-weeks), combined with or in the absence of regular moderate exercise, on cognitive function in a clinical population of older participants identified as experiencing age-related cognitive changes. This project's hypothesis is that the combination of flavonoid-rich diet and routine physical activity may potentiate cognitive benefits and reduce cognitive decline in an aging population, via mechanisms mediated by the gut microbiome.

DETAILED DESCRIPTION:
This randomized clinical trial (RCT) is designed to investigate the effect of 12-weeks blueberry ingestion (50 g freeze dried powder per day, equivalent to 2 cups fresh blueberries per day) with or without brisk walking (five 45-minute supervised sessions per week) on cognitive function in healthy older adult participants. An important aim is to determine if this potential benefit is mediated through changes in the gut microbiome profile and an increase in gut-derived phenolics.

Older adult participants (n=240, with a goal of 200 completing all procedures) will be randomized to one of four groups: blueberry-walking, blueberry-stretching, placebo-walking, and placebo-stretching. The blueberry and placebo powder supplements will be ingested using double blind procedures. Blood, urine, and stool samples will be collected pre-study, and then again after 6- and 12-weeks. Cognitive function and cardiorespiratory fitness will be measured at the same time points. Participants will be assessed for processing speed, episodic memory, working memory, and sustained attention using the Cambridge Neuropsychological Test Assessment Battery (CANTAB, Cambridge Cognition, Ltd) (laboratory of Dr. Carol Cheatham, UNC Chapel Hill). Urine samples will be analyzed for gut-derived phenolic metabolites via liquid chromatography tandem MS/MS (lab of Dr. Mary Ann Lila, NCSU). Taxonomic and functional profiles from metagenomic sequencing of the stool samples will be acquired (UNC Chapel Hill).

Recruitment. Healthy older adult participants (240 to start, 200 to finish) will be recruited from the Charlotte, NC, metropolitan area. Healthy, nonsmoking, physically inactive male and female participants (targeting 65-85 years of age, BMI less than 35) with cognitive changes will be selected who match the inclusion and exclusion criteria.

Design. This study will employ a randomized, double blind, placebo controlled, parallel group research design, with participants (60) assigned to one of 4 arms for the 12 week trial period: blueberry and walking; blueberry and stretching; placebo and walking; placebo and stretching.

Schedule

1. PRE-STUDY SCREENING Before joining the study, potential subjects will participate in a phone call with the research staff (30-60 minutes). We have prepared a phone script for this call. They will receive a brief review of study requirements and then will take the Telephone Interview for Cognitive Status (TICS). The TICS questionnaire is a validated method for use in telephone calls to assess cognition and closely predicts the MoCA score. Only 30% of elderly subjects score within the range acceptable for this study and this prescreening test will help avoid an unnecessary lab visit to the NCRC for 7 of 10 potential subjects. If the test score is within the range that is acceptable for this study, potential subjects will be given further information regarding the study. Study inclusion and exclusion criteria will be reviewed. Three lab visits will be scheduled so that potential subjects can reserve these dates in their calendar. The TICS was specifically developed to be a phone screening instrument. The range of scores on the TICS to determine eligibility for our study is 28-36.

LAB TESTING VISIT #1: Orientation, Consent, and Pre-Study Cognitive and Fitness Testing (approximately 3-4 hours).

A. ORIENTATION AND CONSENT (15 min): Subjects will come to the AppState Human Performance Lab at an assigned time. Study procedures will be thoroughly explained by the research staff during the consent process. Subjects will be invited to voluntarily sign the consent form.

B. COGNITION TESTING, MoCA (5 min): Participants will report to the lab of Dr. Cheatham (UNC Chapel Hill, Nutrition Research Institute, NCRC) where they will undergo cognitive testing using the MoCA. This will confirm the TICS survey taken during the screening phone call. Subjects will be tested for mild cognitive decline using the Montreal Cognitive Assessment (MoCA). The MoCA test consists of eight short sections to test memory, attention, and other similar functions. The MoCA score will be assessed to determine if subjects meet the criteria for mild cognitive decline and thus qualify for this study (24.1-25.2 that indicates mild cognitive decline). Subjects may be excused from further participation in this study depending on the score. Those who score below the 1.5 SD cutoff will be referred to their family physicians.

C. LAB QUESTIONNAIRES AND KITS (15 min): Subjects will complete a physical activity survey and a medical health questionnaire. Subjects will receive a 3-day food record, stool collection kit, and the 24-hour urine collection kit, with complete instructions. The 3-d food record will be completed on the Thursday, Friday, and Saturday period before the first exercise training session. Urine and stool samples will be collected the day before the first exercise training session. The dates/times for additional lab visits will be confirmed. Subjects will receive a log for recording daily step counts with specific instructions.

D. BODY COMPOSITION (10 min): Height and weight will be measured using a stadiometer and balance beam weight scale. The seca medical Body Composition Analyzer (mBCA) (Hanover, MD) will be used to measure body composition through 8 point BIA while participants stand on foot electrodes with bare feet and grasp electrodes with both hands on side rails. The seca mBCA provides several measurements of interest, including fat mass, fat free mass, skeletal muscle mass, visceral fat, total body water, and extracellular water.

E. COGNITION TESTING, CANTAB (45 min): Subjects that qualify for the study using the MoCA criteria will be further tested at Cheatham's lab for cognitive function using the Cambridge Neuropsychological Test Assessment Battery (CANTAB, Cambridge Cognition, Ltd). The CANTAB is a standardized and computerized instrument with automated data capture. Participants will be assessed for processing speed, episodic memory, working memory, and sustained attention. The CANTAB has been validated for assessment of cognitive decline and will be used to validate the findings from the other assessments. The chosen CANTAB collection of subtests (see below) has been designed at Cambridge to assess cognitive decline and has been shown to be sensitive to deterioration of cognitive abilities, even in the short-term. Completion of the 5 subtests requires about 30 minutes. The tasks are completed on a touch screen computer. Subtests of the CANTAB to be included in the battery: Motor Control Task -to familiarize participant with the touch screen; Rapid Visual Information Processing -test of sustained visual attention; Paired Associate Learning -test of memory and learning; Reaction Time -test of simple & choice reaction time; Spatial Working Memory -test of spatial information retention.

F. COGNITION TESTING, ERP (60 min): Subjects will also be assessed using electrophysiological procedures (ERP) in Cheatham's lab. To collect ERP data, the participant will be fitted with a Geodesic Sensor Net (GSN; Electrical Geodesic, Inc.) consisting of a 128-sensor array. The GSN is easy to apply, comfortable, and relatively non-invasive. The GSN is comprised of Ag/AgCl sensors in an elastic-webbed geodesic tension structure. The participant's head is measured to insure the proper net is used and to mark the scalp at the vertex for proper placement of net. The GSN is soaked in a potassium chloride and warm water solution. Excess solution is blotted from the net so that it does not drip in the participant's eyes. The net is carefully stretched over the participant's head matching the vertex electrode to the vertex mark and the ear electrodes with the preauricular points. The chinstrap and side tension straps are tightened and the sensors are all checked to insure that they are perpendicular to and in contact with the scalp. Application of the net requires only about 5 minutes and is well tolerated. A picture will be taken of the net placement and impedances are then checked. Any sensors that are not reading well are adjusted and a small amount of electrolyte solution is applied to the sensor's sponge with a pipette. When impedances are within accepted limits, the participant will be seated in front of the monitor in the participant room (separate from the control room). A camera, which is time-locked to the data being acquired, will record the participant during presentation of the pictures. Using the Smart-Eye eye-tracking system, we will collect information on gaze direction and eyeblinks. This system is the only system on the market to offer integrated dense array EEG and remote head- and eye-tracking for linking attention, time-on-task, pupillometry, and eye blinks to the ongoing EEG. Data will be recorded continuously and epoched into windows around the stimuli presentation offline. Once the net is in place, the participant will participate in the three cognitive tests. For the n-back working memory task, participants will watch a series of letters appearing on the computer screen and will press a button when the target is detected. The target in a 2-back task is identified as a letter that matches the letter that appeared letter-before-last (2-back). Letters that do not match the definition require no response. Use of this task has been shown to predict those in which cognitive decline will be rapid. To assess visual mismatch negativity component of the N200 (attention), the participant will be instructed to focus on the center of the screen. At a ratio of 16:1:1 (standards:targets:deviants), the computer will randomly cycle through the task. When a defined target appears, the participant will press the button. All other stimuli do not require a response. This task requires sharp attentional focus and has been shown to be sensitive to mild cognitive impairment.

G. STRESS QUESTIONNAIRES (10 min): Subjects will complete questionnaires that assess anxiety and stressful life events.

H. BLOOD SAMPLE (5 min): Study participants will return to the AppState Human Performance Lab. Blood samples (maximum of 35 mL) will be collected from an arm vein by a trained phlebotomists while participants are seated.

I. GRADED EXERCISE TREADMILL TEST: Participants will be tested for maximal aerobic capacity (VO2max) during a graded, treadmill test with the Cosmed CPET metabolic cart. Before the test, subjects will be told that they should be rested and hydrated for the test and avoid caffeine and tobacco within 3 hours of testing and avoid alcohol within 12 hours of testing. Subjects will be told to avoid exercising on the day of testing and to report any medication that they are using to the testing staff before the test. Participants will first warm up on the treadmill to demonstrate that they can freely walk on the treadmill. Participants will walk against a gradually increasing workload (Bruce protocol) until maximal effort is reached and the participant voluntarily stops exercising. The main outcome measure is peak VO2 or the milliliters of oxygen that can be consumed for each kilogram of body mass at peak effort. The Cosmed CPET metabolic system (Rome, Italy) will be attached via a facemask to the participant for continuous measurement of metabolic factors (oxygen consumption, ventilation rate, respiratory rate, respiratory exchange ratio). A chest heart rate monitor will provide heart rates in beats per minute. The rating of perceived exertion (RPE) will be assessed using a 6 to 20 scale. Data will be recorded at the end of each 3 minute stage and at the point of maximal exertion, and submaximal/maximal changes pre to post 12 weeks training will be used as criteria for assessing changes in cardiorespiratory fitness. The aerobic exercise prescription for the 12 week training program will be based on the maximal heart rate (MHR) and resting heart rate (RHR) measured during baseline testing. Testing and safety procedures will be under IRB guidance for healthy elderly participants, and the study MD will provide oversight of testing procedures. Subjects that have difficulty in walking on the treadmill and feel they cannot walk for 45 minutes on an outside track will be excused from the research project.

J. SUPPLEMENTS: Each participant will be given a 6-weeks supply of vacuum-sealed packets of coded lyophilized wild blueberry powder or placebo (50 g daily). Subjects will received a handout with specific instructions regarding the supplementation protocol. The lowbush wild blueberry freeze-dried powder will be provided from the Wild Blueberry Association of North America, Old Town, ME and freeze-dried by FutureCeuticals (Momence, IL). The fiber and carbohydrate-matched placebo blueberry powder will be developed by NCSU using a formula from previous studies: blueberry flavoring and aroma (8.9%), coloring (1.05% purple lake, 0.75% red lake, 0.45% blue 2 lake, 0.03% red dye, 0.008% blue 2 dye), glucose (32%), fructose (35.5%), citric acid (0.77%), cellulose (15%), fibersol-2 (1.8%), xanthan gum (1%), pectin (1.09%) and silica (0.99%). The blueberry and placebo powders will be packaged at the NCRC NC Food Innovation Lab. Participants will be instructed that the blueberry or placebo powders should be stored in a freezer in the supplied packets until use. Instructions will be provided to consume the supplements in split doses (half with breakfast and half with lunch) mixed in beverages, yogurt, or other foods. If a study participant fails to take the supplement dose on a given day or two, they will be asked to add 1 extra packet per day until they are back on schedule. Study participants will contact the Research Manager (ASU-NCRC@appstate.edu) if they fail to consume the supplement for 3 days or longer, and discuss whether or not they wish to dropout of the study. Compliance to the supplementation regimen will be assessed through regular email messages and a count of returned packets at the 6- and 12-week time points.

LAB TESTING VISITS #2 and #3. These same basic procedures will be repeated after 6- and 12-weeks except that visits #2 and #3 will not involve going through the consent process and completing the medical health questionnaire, and that visit #3 will not include providing additional supplement packets. Study participants will be asked if any change has occurred in their health status since the previous visit. If adherence to the inclusion and exclusion criteria have changed, this will be reviewed with the study participant.

12-WEEK RANDOMIZED CLINICAL TRIAL: 60 TRAINING SESSIONS AT THE NORTH CAROLINA RESEARCH CAMPUS (NCRC, Kannapolis, NC)

* Participants will engage in supervised physical activity sessions (5 SESSIONS PER WEEK, 45 MIN PER SESSION) and consume 50 grams per day of freeze-dried blueberry powder or placebo.
* Participants will engage in 45 minutes per day supervised exercise (brisk walking with heart rate monitors, or non aerobic stretching floor exercises) for 5 days per week during a 12-week period. Exercise sessions will be conducted in small groups under supervision. Exercise supervisors will be trained in CPR, and an AED device will be located at the door of the Human Performance Lab (in the building adjacent to the walking oval).
* Walking sessions will be held outdoors under supervision on the NCRC track. Training heart rates and total distance walked will be recorded. On days with inclement weather, subjects will walk under cover (NCRC parking garage) or on treadmills in the Human Performance Lab.
* Heart rate during the physical activity sessions will be monitored with a FitBit Inspire. Walkers will gradually increase intensity with a goal of 60% of the heart rate reserve (based on data from the graded exercise test).
* The stretching program will be supervised and conducted in the Human Performance Lab on mats. The session will start with 5 to 10 minutes warm up of light activity (e.g., easy walking with light calisthenics). After the warm up, participants will engage in 8 to 10 stretching exercises per session under the guidance of an exercise supervisor. Each stretching exercise will be held for 10 to 30 seconds at the point of slight discomfort. The flexibility exercise will be repeated for two to four repetitions, with participants aiming for 60 seconds of total stretching time per flexibility exercise (e.g., four 15 second stretches). Exercise supervisors will provide a complete orientation to the stretching exercises during the first session.
* All subjects will record total daily step counts (from when they get out of bed in the morning until getting into bed to sleep in the evening) from the Fitbit just before bedtime each day of the study. Subjects will be instructed to take the FitBit off during sleep and put it back on their wrist when awakening. Subjects will charge the FitBit on a weekly basis.
* Two primary cohorts (40 each, walking and stretching groups) will be scheduled each semester during a 3-month period (September through November, and February through April) during a 3-year period. Of 240 participants entered into the study each year, 200 are expected to successfully complete all phases. Retention will be maximized by regular contact with participants during supervised exercise sessions and through regular email messages. Two exercise session times will be offered each day of the work week (approximately 8:00 am and 2:00 pm). If participants miss an exercise session, there will be weekly opportunities to attend make up sessions (Saturday mornings). Study participants will be allowed an average of one exercise session per week to be unsupervised (e.g., during out-of-town travel, holidays, etc.). If a study participant misses 3 or more days of exercise training, the Research Manager will contact the participant and discuss whether or not they want to drop out of the study.

ELIGIBILITY:
Inclusion Criteria:

* Score on the Montreal Cognitive Assessment (MoCA test) of 24.1-25.2 that indicates mild cognitive decline. The MoCA test score ranges from 0 to 30, with higher scores from 26 to 30 considered normal.
* Healthy, non-smoking male or female participants 65 to 85 years of age.
* Capable of engaging in a supervised 12-week exercise training program (brisk walking or stretching).
* Physically inactive (defined as less than 150 min/week moderate or less than 75 minutes vigorous aerobic and/or resistance exercise during the past 4 weeks).
* Willingness to be randomized to one of four groups.
* Willingness to provide blood, urine, and fecal samples (3 each),
* Willingness to avoid blueberry intake during the 12-weeks study (other than what is provided through the study).
* Willingness to maintain current diet and physical activity patterns during the study (other than what is prescribed as a part of the study), and make no formal attempts to lose or gain body weight.
* Willingness to be a participant in this study only and not enter any other studies.

Exclusion Criteria:

* Allergy to blueberries.
* Diagnosis of Type I or Type 2 diabetes.
* Chronic cardiovascular, metabolic, or renal condition that is uncontrolled (controlled defined as stable for 6 months or more).
* History of signs or symptoms during rest or physical activity such as chest discomfort, unreasonable breathlessness, dizziness, fainting, or blackouts.
* Use of any prescription or over-the-counter drug intended to support cognition or with known cognitive side effects.
* Any other concurrent condition or use of medications or supplements which, in the opinion of the study clinician would preclude participation in this study.
* Diagnosis of dementia.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognition | Change from pre-study to 6-weeks and 12-weeks
  Cognitive function using the Cambridge Neuropsychological Test Assessment Battery (CANTAB, Cambridge Cognition, Ltd).

SECONDARY OUTCOMES:
Maximal aerobic capacity | Change from pre-study to 6-weeks and 12-weeks
  VO2max from a graded treadmill test using a metabolic cart
Gut microbiome | Change from pre-study to 6-weeks and 12-weeks
  Alpha and beta diversity from gut microbiome taxa analysis using Whole Genome Shotgun (WGS) sequencing
Urine blueberry metabolites | Change from pre-study to 6-weeks and 12-weeks
  Urine gut-derived metabolites (n=24) from targeted LC-MS/MS analysis (concentrations) generated from blueberry ingestion
Electrophysiological procedures (ERP) using the Geodesic Sensor Net | Change from pre-study to 6-weeks and 12-weeks
  An electroencephalogram (EEG) test that measures cognition from electrical activity (amplitude in microvolts) in the brain in response to cognitive challenges including working memory

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When the study is completed in 2028 and will be available for five years afterwards.
Access Criteria: Researchers with relevant expertise and a track record in the research area related to the IPD can request access.
  Researchers must submit a research proposal outlining their research goals, analysis plan, and how the IPD will be used.